CLINICAL TRIAL: NCT04311931
Title: The Effect of a Creative Dance Program on Well-being, Physical Function, Body Awareness, and Rhythm Perception and Reproduction of Community-dwelling Older Adults
Brief Title: Creative Dance Effects on Community-dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Collaborators: Departamento de Desporto e Saúde, Escola de Ciências e Tecnologia, Universidade de Évora, Évora, Portugal (Unknown); Comprehensive Health Research Center (Other); Horizon 2020 - Portugal 2020 (ALT20-03-0145-FEDER-000007 - Project: ESACA) (Unknown)
Responsible Party: Principal Investigator, Ana Cruz-Ferreira, Principal Investigator, University of Évora
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UEvora Dance 2020
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Community-dwelling Older Adults
Keywords: Older adults; Creative dance; Well-being; Life satisfaction; Affects; Physical function; Body awareness; Rhythm
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Creative Dance group (Experimental): The experimental group intervention will attend the creative dance program. The program integrates 3 sessions / week of 60 minutes on alternated days.
  Interventions: Other: Active Dance Program
- Control group (No Intervention): The control group will maintain the usually daily activities, not attending any exercise program.
  After study end, the control group will have the opportunity to participate on an exercise program.

INTERVENTIONS:
Other: Active Dance Program — All Creative Dance sessions comprised five phases: 1) opening ritual (5 min), in which participants will be welcomed and will be informed about the objectives and structure of the session; 2) warm-up (15 min), in which body muscle groups will be activated through the introduction of basics elements of movement; 3) main phase (30 min), will be proposed individual, pair and group activities, in order to achieve the objectives described above. This phase will end with a choreography composition; 4) cool-down (5 min) with stretching and physiological parameters normalization; and 5) ending ritual (5 min), in which the participants will be invented to share their sessions' experience and they will fill a sheet with attendance, exercise intensity perception (Borg Scale) and satisfaction's (Caregiver Treatment Satisfaction questionnaire).
  Arms: Experimental Creative Dance group

SUMMARY:
The aim of present study is to analyze the effect of a Creative Dance program on well-being, physical function, body awareness, and rhythm perception and reproduction of community-dwelling older adults. This quasi-experimental study is a controlled trial.

Participants will be allocated to two groups: experimental group (who attend the Creative Dance program) and control group (who maintain usual activity).

The Creative Dance program will run for 12 weeks (3 sessions/week of 60 minutes).

Participants will be assessed 1) at baseline and at 2) at 12 weeks.

DETAILED DESCRIPTION:
An healthspan life obey older adults to adhere to an active ageing lifestyle because it combat the natural cognitive and physical losses associated with ageing (1-3). Exercise programs have shown to be effective interventions for healthspan (2) and its attendance is high recommended by health organizations (4). Several studies have analyzed the beneficial effects of exercise programs on physical and cognitive performance of older adults, and they concluded that multimodal programs involving both physical and cognitive stimulation are more benefic than single physical or cognitive program interventions (5). Dance involves both physical and cognitive stimulation, since the participants are engaged physical, intellectually, and emotionally tasks(6). Dance explore the movement elements (body, space, time, dynamic, and relationships) and particularly the Creative Dance explore it through tasks that allow the participants to create their own movements and express ideas and feelings through body language (7). In Creative dance, tasks can be simplified according to specificities/limitations of participants and considering a holist approach (6). This dance do not require any dance technique or prior training, and promote socioemotional interactions, stimulating positive feelings, joy, and pleasure; furthermore, is a safe practice, not requiring expensive resources (6). For these reasons, Creative Dance is becoming gradually recommended for older people by investigators (6-9). In fact, Creative Dance seems to increase proprioception (8), several physical fitness parameters (7, 9), mobility (9) and life satisfaction (7) of older people. Thus, although there are only few studies in Creative Dance for older adults, this form of dance seems to be a pertinent practice to revert their usual process of loss and decline of motor and mental skills (6). We hypnotized, that a Creative Dance program may contribute to the community-dwelling older adults' healthspan, particularly we hypnotized that such program may induce improvements on physical fitness, on body awareness, and on rhythm perception and reproduction, as well to promote improvements on well-being indicators.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥60 years;
* Community-dwelling older adults living independently.

Exclusion Criteria:

* Presence of cognitive impairment (Mini-Mental State Examination) (11);
* Presence of motor impairment, neurological problems or diseases compromising the program participation;
* Participation in regular physical exercise during the previous 6 months;
* Unavailability to participate in the program.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Life satisfaction | [ 0, 12 weeks]
  Change from Baseline, between and within groups comparison, in well-being outcome measure Life Satisfaction assessed by Satisfaction With Life Scale, ranging from 5 (worst) to 25 (best) points (10), Portuguese version (11).
Affects | [ 0, 12 weeks]
  Change from Baseline, between and within groups comparison, in well-being outcome measure Positive Affects assessed by Positive and Negative Affect Schedule (PANAS), ranging from 10 (worst) to 50 (best) points (12), Portuguese version (13).
Affects | [ 0, 12 weeks]
  Change from Baseline, between and within groups comparison, in well-being outcome measure Negative Affects assessed by Positive and Negative Affect Schedule (PANAS), ranging from 10 (best) to 50 (worst) points (12), Portuguese version (13).
Depressive Status | [ 0, 12 weeks]
  Change from Baseline, between and within groups comparison, in well-being outcome measure Depressive Status assessed by the Short Form of Geriatric Depression Scale, ranging from 0 (best) to 15 (worst) points (14), Portuguese version (15).
Balance | [ 0, 12 weeks]
  Change from Baseline, between and within groups comparison, in Physical Fitness outcome measure Balance assessed by the Fullerton Advanced Balance Scale, ranging from 0 (worst) to 40 (best) points (16, 17).
Agility | [ 0, 12 weeks]
  Change from Baseline, between and within groups comparison, in Physical Fitness outcome measure Agility and Balance assessed by Timed Up and Go test (18).
Coordination | [ 0, 12 weeks]
  Change from Baseline, between and within groups comparison, in Physical Fitness outcome measure Coordination assessed by an adapted form for older adults of the "Rhythm Test de Evaluación de la Habilidad Motora" from Ortega and Blázquez, ranging from 3 (worst) to 12 (best) points (19) while counting backward by one from 100.
Rhythm perception and reproduction | [ 0, 12 weeks]
  Change from Baseline, between and within groups comparison, in rhythm perception and reproduction assessed by an adapted form for older adults of the "Rhythm Test of Batterie d'évaluations des fonctions neuro-psychomotrices", ranging from 0 (worst) to 6 (best) points (20)(21).
Body Awareness | [ 0, 12 weeks]
  Change from Baseline, between and within groups comparison, in Body Awareness assessed by the Multidimensional Assessment of Interoceptive Awareness (22), ranging from 0 (worst) to 165 (best) points, Portuguese version (23).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Cruz-Ferreira, PhD, Principal Investigator — University of Évora
Locations (1):
- Ana Cruz-Ferreira, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crimmins EM. Lifespan and Healthspan: Past, Present, and Promise. Gerontologist. 2015 Dec;55(6):901-11. doi: 10.1093/geront/gnv130. Epub 2015 Nov 10. PMID 26561272
- [Background] Berthelot G, Johnson S, Noirez P, Antero J, Marck A, Desgorces FD, Pifferi F, Carter PA, Spedding M, Manoux AS, Toussaint JF. The age-performance relationship in the general population and strategies to delay age related decline in performance. Arch Public Health. 2019 Dec 9;77:51. doi: 10.1186/s13690-019-0375-8. eCollection 2019. PMID 31827790
- [Background] Berthelot G, Bar-Hen A, Marck A, Foulonneau V, Douady S, Noirez P, Zablocki-Thomas PB, da Silva Antero J, Carter PA, Di Meglio JM, Toussaint JF. An integrative modeling approach to the age-performance relationship in mammals at the cellular scale. Sci Rep. 2019 Jan 23;9(1):418. doi: 10.1038/s41598-018-36707-3. PMID 30674921
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Levin O, Netz Y, Ziv G. The beneficial effects of different types of exercise interventions on motor and cognitive functions in older age: a systematic review. Eur Rev Aging Phys Act. 2017 Dec 21;14:20. doi: 10.1186/s11556-017-0189-z. eCollection 2017. PMID 29276545
- [Background] Cruz-Ferreira A, Alves MJ, Pereira C. A Dança: uma prática para a pessoa idosa. In: Mendes, F., Pereira, C., & Bravo, J. (Ed. UÉ). Envelhecer em Segurança no Alentejo. Compreender para agir. ISBN: 978-989-99122-9-8. Évora, PT. In: Mendes F, Pereira C, Bravo J, editors. Envelhecer em Segurança no Alentejo Compreender para agir. Évora: Universidade de Évora; 2020.
- [Background] Cruz-Ferreira A, Marmeleira J, Formigo A, Gomes D, Fernandes J. Creative Dance Improves Physical Fitness and Life Satisfaction in Older Women. Res Aging. 2015 Nov;37(8):837-55. doi: 10.1177/0164027514568103. Epub 2015 Jan 29. PMID 25651595
- [Background] Marmeleira JF, Pereira C, Cruz-Ferreira A, Fretes V, Pisco R, Fernandes OM. Creative dance can enhance proprioception in older adults. J Sports Med Phys Fitness. 2009 Dec;49(4):480-5. PMID 20087310
- [Background] Joung HJ, Lee Y. Effect of Creative Dance on Fitness, Functional Balance, and Mobility Control in the Elderly. Gerontology. 2019;65(5):537-546. doi: 10.1159/000499402. Epub 2019 May 3. PMID 31055579
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Simões A. Ulterior validação de uma escla de satisfação com a vida. Revista Portuguesa de Pedagogia. 1992;26:503-15.
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Galinha I, Pereira C, Esteves F. Versão reduzida da escala portuguesa de afeto positivo e negativo - PANAS - VRP: Análise fatorial confirmatória e invariância temporal. Psicologia. 2014;28(1):50-62.
- [Background] Yesavage JA, Sheikh JI. 9/Geriatric depression scale (GDS) recent evidence and development of a shorter version. Clinical gerontologist. 1986;5(1-2):165-73.
- [Background] Apóstolo J, Loureiro L, Reis I, Silva I, Cardoso D, Sfetcu. R. Contribuição para a adaptação da Geriatric Depression Scale -15 para a língua portuguesa. Revista de Enfermagem Referência. 2014;20(3):65-73.
- [Background] Pereira C, Baptista F, Cruz-Ferreira A. Role of physical activity, physical fitness, and chronic health conditions on the physical independence of community-dwelling older adults over a 5-year period. Arch Gerontol Geriatr. 2016 Jul-Aug;65:45-53. doi: 10.1016/j.archger.2016.02.004. Epub 2016 Feb 17. PMID 26966842
- [Background] Hernandez D, Rose DJ. Predicting which older adults will or will not fall using the Fullerton Advanced Balance scale. Arch Phys Med Rehabil. 2008 Dec;89(12):2309-15. doi: 10.1016/j.apmr.2008.05.020. Epub 2008 Nov 1. PMID 18976981
- [Background] Rikli RE, Jones CJ. Development and validation of criterion-referenced clinically relevant fitness standards for maintaining physical independence in later years. Gerontologist. 2013 Apr;53(2):255-67. doi: 10.1093/geront/gns071. Epub 2012 May 20. PMID 22613940
- [Background] Domingues D. Psicomotricidad e intervención educativa: Psicologia Pirámide; 2008.
- [Background] Vaivre-Douret L. NP-MOT - Batterie d'Évaluations des Fonctions Neuro-Psychomotrices de l'enfant. Appliquée. LEdCdP, editor. Paris2006.
- [Background] Vaivre-Douret L. Batterie d'évaluations des fonctions neuro-psychomotrices de l'enfant. Le Carnet PSY. 2007;2(115):27.
- [Background] Mehling WE, Price C, Daubenmier JJ, Acree M, Bartmess E, Stewart A. The Multidimensional Assessment of Interoceptive Awareness (MAIA). PLoS One. 2012;7(11):e48230. doi: 10.1371/journal.pone.0048230. Epub 2012 Nov 1. PMID 23133619
- [Background] Machorrinho J, Veiga G, Fernandes J, Mehling W, Marmeleira J. Multidimensional Assessment of Interoceptive Awareness: Psychometric Properties of the Portuguese Version. Percept Mot Skills. 2019 Feb;126(1):87-105. doi: 10.1177/0031512518813231. Epub 2018 Nov 19. PMID 30451581
- [Derived] Rosado H, Motta P, Almeida G, Cruz-Ferreira A, Pereira C. Exploring the benefits of a psychomotor intervention mediated by creative dance in community-dwelling older adults: development of new coordination and rhythm tests. BMC Public Health. 2025 May 14;25(1):1780. doi: 10.1186/s12889-025-21478-0. PMID 40369447